CLINICAL TRIAL: NCT03809273
Title: Effects of Yangxinshi Pills on the Exercise Tolerance Compared With Trimetazidine in Patients After PCI: a Prospective，Muhicenter,Doubleblind, Double-dummy, Randomized, Controlled Trial
Brief Title: Effects of Yangxinshi Pills on the Exercise Tolerance Compared With Trimetazidine in Patients After PCI
Acronym: HEARTRIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Director, clinical professor, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GrowfulPower-001
Record Dates: First submitted 2019-01-03; First posted 2019-01-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Cardiopulmonary Exercise Test
MeSH Terms: interventions — Yangxinshi; Trimetazidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yangxinshi (Experimental)
  Interventions: Drug: Yangxinshi; Drug: Trimetazidine mimic
- Trimetazidine (Active Comparator)
  Interventions: Drug: Trimetazidine; Drug: Yangxinshi mimic

INTERVENTIONS:
Drug: Yangxinshi — Yangxinshi pill 3 pills /tid
  Arms: Yangxinshi
Drug: Trimetazidine — Trimetazidine 20mg/tid
  Arms: Trimetazidine
Drug: Yangxinshi mimic — Yangxinshi mimic tablets 3 pills /tid
  Arms: Trimetazidine
Drug: Trimetazidine mimic — Trimetazidine mimic tablets 20mg/tid
  Arms: Yangxinshi

SUMMARY:
This study compared the effect of Yangxinshi on exercise tolerance of patients with percutaneous coronary intervention (PCI) for the first time with Trimetazidine.Half of participants will receive Yangxinshi and Trimetazidine mimic tablets in combination,While the other half will receive Trimetazidine and Yangxinshi mimic tablets.

DETAILED DESCRIPTION:
The Primary Purpose of this study is to compare the effect of Yangxinshi on exercise tolerance of patients with percutaneous coronary intervention (PCI) for the first time with Trimetazidine, The target patients are the people who underwent PCI for the first time and can be carried on Cardiopulmonary exercise test. The treatment period was 24 weeks. The patients were randomly divided into two groups.： A: Yangxinshi pill 3 pills /tid and Trimetazidine mimic tablets 20mg/tid B: Trimetazidine mimic tablets 20mg/tid and Yangxinshi pill 3 pills /tid The patients were followed up for 0 weeks, 4 weeks, 12 weeks, 24 weeks and 28 weeks after entering the group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~ 75, gender is not limited；
* The patient within two month after PCI operation for the first time；
* The patient had 1-2 coronary artery lesions with complete revascularization：At least one drug eluting stent was implanted，and residual coronary artery stenosis after PCI <30%；
* Have not revascularization plan within 6 months；
* After being evaluated by clinicians on aerobic exercise ability，patients can carry out early rehabilitation in hospital and exercise cardiopulmonary rehabilitation outside the hospital；
* Coronary heart disease patients with Qi Deficiency and Blood Stasis Syndrome；
* Participants voluntarily participated in and signed informed consent；

Exclusion Criteria:

* Patients was diagnosed with AMI as the first diagnosis in the past month, and then hospitalized for PCI operation；
* Patients with absolute and relative contraindications in cardiopulmonary exercise test；
* Any drug allergy to Yangxinshi pill and trimetazidine；
* Patients have taken regular Yangxinshi pill, trimetazidine or other Chinese patent medicine regularly in the past month；
* Patients are intolerant of aspirin, clopidogrel, statins, beta blockers or ACEI drugs (such as massive hemorrhage, severe hypotension, etc.)；
* History of stroke (cerebral hemorrhage, subarachnoid hemorrhage, cerebral thrombosis, cerebral embolism and stroke of unknown type) or lower extremity arterial disease in the past 6 months
* Active bleeding disease within 6 months；
* Combined with severe liver and kidney dysfunction (creatinine clearance ≤ 30ml / min or in the active stage of kidney disease, serum aminotransferase ≥ 3 × upper limit of clinical reference), other lifethreatening serious primary or psychiatric diseases and malignant tumors
* Hemoglobin <90 g/L；
* Cardiac function (NYHA) grade IV or echocardiography LVEF < 30%；
* Venous blood pressure <100/60 mmHg；
* In past 6 months, have medical history of: pregnancy, prepare or suspected of pregnancy, abortion, breastfeeding or after childbirth
* The expected survival period is less than one year.；
* Patients who are participating in other clinical studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 681 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in METs assessed by the CPET | 24 weeks
  MET=Metabolic Equivalent of Task; CPET=Cardiopulmonary Exercise Test

SECONDARY OUTCOMES:
Changes of anaerobic threshold (AT) by CPET | 24 weeks
Incidence of major cardiovascular events (MACE) | 4,12,24 and 28 weeks
PHQ-9 Depression Scale | 24 weeks
  PHQ=Patient health questionaire, score range: 0-27
Changes of Seattle Angina Questionnaire | 24 weeks
  The Seattle Angina Questionaire (SAQ) quantifies patients'physical limitations caused by angina. The scale is transformed to a score of 0 to 100, where higher scores indicate better function (less physical limitation)
Frequency of angina pectoris | 24 weeks
The proportion of METs>7 patients | 24 weeks
  MET=Metabolic Equivalent of Task
Changes of VO2max by CPET | 24 weeks
Changes of VO2/HR by CPET | 24 weeks
Changes of VO2/W by CPET | 24 weeks
GAD-7 Anxiety Screening Scale | 24 weeks
  GAD=Generalized Anxiety Disorder, score range: 0~21

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Changchun Traditional Medicine University Affiliated Hospital, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Li Y, Zhang Z, Zhang J, Chen H, Yu H, Meng X, Yuan H, Shao L, Lu Y, Liu B, Xu J, Zhang Y, Li J, Han Y; HEARTRIP investigators. Efficacy and safety of yangxinshi versus trimetazidine on exercise tolerance in patients with coronary heart disease after percutaneous coronary intervention: Multicenter, double-blind clinical trial. Phytomedicine. 2024 Dec;135:156198. doi: 10.1016/j.phymed.2024.156198. Epub 2024 Nov 7. PMID 39566404